CLINICAL TRIAL: NCT00706134
Title: An Eight-week Double-blind, Multi-center, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Aliskiren 75 mg, 150 mg, and 300 mg in Elderly Patients With Essential Hypertension When Given With a Light Meal
Brief Title: Efficacy and Safety of Aliskiren 75 mg, 150 mg, and 300 mg in Elderly Patients With Essential Hypertension When Given With a Light Meal in a 8 Week Placebo-controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2405
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Hypertension; ≥ 65 years; aliskiren; placebo; light meal
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Aliskiren 75 mg (Experimental)
  Interventions: Drug: Aliskiren 75 mg
- Aliskiren 150 mg (Experimental)
  Interventions: Drug: Aliskiren 150 mg
- Aliskiren 300 mg (Experimental)
  Interventions: Drug: Aliskiren 300 mg

INTERVENTIONS:
Drug: Placebo — Placebo tablet taken once daily in the morning with a light meal.
  Arms: Placebo
Drug: Aliskiren 75 mg — Aliskiren 75 mg tablet taken once daily in the morning with a light meal.
  Arms: Aliskiren 75 mg
Drug: Aliskiren 150 mg — Aliskiren 150 mg tablet taken once daily in the morning with a light meal.
  Arms: Aliskiren 150 mg
Drug: Aliskiren 300 mg — Aliskiren 300 mg tablet taken once daily in the morning with a light meal.
  Arms: Aliskiren 300 mg

SUMMARY:
This study will evaluate the efficacy and safety of aliskiren 75 mg, 150 mg, and 300 mg in elderly patients with essential hypertension when given with a light meal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 65 years of age and older.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).
* At the randomization visit patients must have an office msSBP greater than or equal to 150 mmHg and < 180 mmHg (msDBP <110 mmHg) with a less than or equal to 15 mmHg difference during the last two visits of the single blind run-in period.

Exclusion Criteria:

* Severe hypertension [Office msDBP ≥110 mmHg and/or mean sitting systolic blood pressure (msSBP) ≥ 180 mmHg].
* History or evidence of a secondary form of hypertension.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy or cerebrovascular accident, including a history of transient ischemic cerebral attack (TIA).
* Current diagnosis of heart failure (NYHA Class II-IV).
* History of myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI).
* Current angina pectoris requiring pharmacological therapy other than nitrates.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 756 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Investigative Site, Buenos Aires, Argentina
- Investigative Site, Prague, Czechia
- Investigative Site, Berlin, Germany
- Investigative Site, Reykjavik, Iceland
- Investigative Site, Rome, Italy
- Investigative Site, Amsterdam, Netherlands
- Investigative Site, Warsaw, Poland
- Investigative Site, Bratislava, Slovakia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Started | 189 | 192 | 189 | 186
Entered Double-blind Period | 187 | 192 | 189 | 186
Completed | 169 | 173 | 183 | 175
Not Completed | 20 | 19 | 6 | 11
Not completed — Adverse Event | 8 | 7 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 6 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 9 | 3 | 3 | 5
Not completed — Did not meet study criteria | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg | Total
Number analyzed (Participants) | 189 | 192 | 189 | 186 | 756
Age, Customized [Number; unit: Participants]
  ≥ 65 and < 75 years of age | 128 | 131 | 129 | 129 | 517
  ≥ 75 years of age | 61 | 61 | 60 | 57 | 239
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 109 | 106 | 102 | 417
  Male | 89 | 83 | 83 | 84 | 339

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP)From Baseline to End of Study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: Full analysis set (FAS) - All randomized patients. Two randomized patients who did not meet study criteria were excluded from the FAS.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 184 | 192 | 188 | 186
mmHg | -7.97 (1.043) | -12.51 (1.024) | -15.28 (1.035) | -14.14 (1.042)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 184 | 192 | 188 | 186
mmHg | -3.50 (0.579) | -5.33 (0.568) | -6.42 (0.575) | -6.66 (0.579)

3. Secondary Outcome: Percentage of Patients Achieving Systolic Blood Pressure Response
Description: Patients achieving a systolic blood pressure response had to have a msSBP < 140 mmHg at the end of the study and/or a ≥ 20 mmHg reduction in msSBP from baseline to the end of the study.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 184 | 192 | 188 | 186
Percentage of participants | 28.8 | 42.4 | 44.1 | 47.3

4. Secondary Outcome: Change in Mean 24 Hour Ambulatory Systolic and Diastolic Blood Pressure From Baseline to End of Study
Description: Two 24-hour ambulatory blood pressure monitoring (ABPM) evaluations were performed, one at baseline and one at the end of the study. For each evaluation, the ABPM device was attached to the non-dominant arm of the patient.
Time Frame: Baseline to end of study (Week 8)
Population: Ambulatory blood pressure monitoring completers population: All patients that completed both ambulatory blood pressure monitoring assessments successfully.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 50 | 64 | 70 | 58
mmHg
  Ambulatory Systolic Blood Pressure | -1.15 (1.280) | -3.33 (1.155) | -5.76 (1.128) | -5.83 (1.520)
  Ambulatory Diastolic Blood Pressure | 0.31 (0.990) | -1.78 (0.877) | -3.26 (0.693) | -2.45 (0.823)

5. Secondary Outcome: Change in the Smoothness Index (SI) of the Ambulatory Systolic Blood Pressure From Baseline to End of Study (Week 8)
Description: Smoothness index (SI) is a measure of consistency of the BP reduction over 24 hours. The SI was obtained by first calculating the mean blood pressure value at each hour of the 24-hour ambulatory blood pressure monitoring period, both before and during treatment. Similarly, the change from baseline in blood pressure was calculated at each hour. The average hourly change from baseline (δh) and standard deviation (std δh) of the hourly changes were computed, and the SI was derived: SI = δh/std δh. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 50 | 64 | 70 | 58
Ratio | -0.11 (0.102) | -0.38 (0.092) | -0.50 (0.089) | -0.51 (0.096)

6. Secondary Outcome: Change in Morning Surge of Ambulatory Systolic Blood Pressure From Baseline to End of Study (Week 8)
Description: The morning surge was defined as the average of the hourly means in the last three hours (hours 22, 23, 24) of the 24 hour ambulatory blood pressure monitoring assessment period.
Time Frame: Baseline to end of study (week 8)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Number analyzed (Participants) | 50 | 64 | 70 | 58
mmHg | 0.46 (1.782) | -3.04 (1.596) | -7.03 (1.539) | -3.96 (1.660)

ADVERSE EVENTS:
Time Frame: End of study (week 8)
Description: Population description of safety set.
Arm/Group | Placebo | Aliskiren 75 mg | Aliskiren 150 mg | Aliskiren 300 mg
Serious Adverse Events (participants affected / at risk) | 1/186 | 2/191 | 3/189 | 0/188
Other Adverse Events (participants affected / at risk) | 0/186 | 0/191 | 0/189 | 0/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Aliskiren 75 mg (N=191) | Aliskiren 150 mg (N=189) | Aliskiren 300 mg (N=188)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.